CLINICAL TRIAL: NCT03558737
Title: Nasal High-frequency Jet Ventilation (nHFJV) Following Extubation in Preterm Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to safety reasons.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Bradley Yoder, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109858
Record Dates: First submitted 2018-04-25; First posted 2018-06-15 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Infant,Premature; Respiratory Failure; Respiratory Insufficiency; Respiratory Distress Syndrome in Premature Infant
Keywords: non-invasive high frequency ventilation (nHFJV); nasal intermittent positive pressure ventilation (NIPPV)
MeSH Terms: conditions — Premature Birth; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Infants will be stratified by GA (24 0/7 to 25 6/7, 26 0/7 to 28 6/7) and randomized to either nHFJV or NIPPV
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal high-frequency jet ventilation (nHFJV) (Active Comparator)
  Interventions: Other: Nasal high-frequency jet ventilation (nHFJV)
- Nasal intermittent positive pressure ventilation (NIPPV) (Active Comparator)
  Interventions: Other: Nasal intermittent positive pressure ventilation (NIPPV)

INTERVENTIONS:
Other: Nasal high-frequency jet ventilation (nHFJV) — Non-invasive high-frequency jet ventilation provided via the Bunnell Life Pulse high-frequency JET ventilator through a Rusch latex nasopharyngeal airway
  Arms: Nasal high-frequency jet ventilation (nHFJV)
Other: Nasal intermittent positive pressure ventilation (NIPPV) — Non-invasive positive pressure ventilation delivered via a conventional ventilator through Hudson prongs
  Arms: Nasal intermittent positive pressure ventilation (NIPPV)

SUMMARY:
Very low birth weight infants are at increased risk of requiring prolonged duration of mechanical ventilation and multiple intubations, both of which are risk factors for ventilator-induced lung injury and BPD. Thus, it is important to investigate respiratory support methods that are able to effectively oxygenate and ventilate these high risk preterm infants while reducing their risk of lung injury. Nasal high-frequency ventilation is one potential intervention that may decrease the risk of respiratory failure in very low birth weight infants. Small studies have shown effective respiratory support over short time periods in infants, however these studies use nasal high-frequency oscillatory ventilation. To the investigators' knowledge there is no published studies looking at the use of nasal high-frequency jet ventilation in this high risk population.

Use of non-invasive high frequency ventilation (HFV) has been described as a rescue method following failure of other non-invasive ventilator modes or as a means to increase the success post-extubation. When used as invasive high frequency ventilation, high frequency oscillatory ventilation (HFOV) or high frequency jet ventilation (HFJV) utilize supraphysiologic respiratory rates and small tidal volumes which has been shown to inflict less lung injury than conventional modes of ventilation.

Using a mechanical newborn lung model, nasal HFV has improved CO2 removal when compared to conventional NIPPV. Animal studies in the lab of Kurt Albertine have shown improved ventilation and oxygenation in the high frequency nasal ventilation group versus the mechanical ventilation group in a preterm lamb model leading towards better alveolar formation noted histologically.

The investigators hypothesize that extubation of very preterm infants to nHFJV will significantly decrease the rates of reintubation compared to those infants extubated to NIPPV.

ELIGIBILITY:
Inclusion Criteria:

* 24 0/7 to 28 6/7 weeks GA
* Intubated within 24 hours of life to synchronized intermittent mandatory ventilation (SIMV) or high frequency ventilation (HFV, includes HFOV or HFJV)
* Plan for extubation within 72 hours of life
* Infants intubated for surfactant replacement therapy via INSURE method (Intubation-Surfactant-Extubation) are eligible
* Consent obtained from parent/legal guardian

Exclusion Criteria:

* Major congenital and/or chromosomal anomalies
* Upper oropharyngeal anomalies

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Yoder, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated after only 2 subjects enrolled in each arm.
Period: Overall Study
Arm/Group | Nasal High-frequency Jet Ventilation (nHFJV) | Nasal Intermittent Positive Pressure Ventilation (NIPPV)
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Babies born between 24 weeks and 28 weeks completed gestation were screened for enrollment. This study was terminated early and enrolled three 25 week GA infants and one 28 week GA infant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal High-frequency Jet Ventilation (nHFJV) | Nasal Intermittent Positive Pressure Ventilation (NIPPV) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Customized [Mean (Full Range); unit: Weeks] — Completed weeks gestation at delivery
  Weeks
    GA at delivery | 26.5 [25 to 28] | 25 [25 to 25] | 25.75 [25 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: 72 Hour Rate of Reintubation to Invasive Mechanical Ventilation
Description: The number of participants who needed to be reintubated during the first 72 hours of initiation of study intervention will be compared between both arms.
Time Frame: 72 hours
Population: 2 participants were randomized to each arm. All of the participants required reintubation during the initial 72 hour treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal High-frequency Jet Ventilation (nHFJV) | Nasal Intermittent Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

2. Secondary Outcome: Rates of Moderate to Severe Bronchopulmonary Dysplasia (BPD)
Description: The number of infants diagnosed with moderate to severe BPD evaluated at 36 weeks corrected gestational age as defined by the 2001 NICHD Consensus Conference, with and without altitude correction will be compared between both arms
Time Frame: 6 to 12 weeks
Population: One infant in each group had died prior to the evaluation for BPD.
Measure: Number; unit: number participants diagnosed with BPD
Arm/Group | Nasal High-frequency Jet Ventilation (nHFJV) | Nasal Intermittent Positive Pressure Ventilation (NIPPV)
Number analyzed (Participants) | 1 | 1
number participants diagnosed with BPD | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events collected from placement on nasal respiratory support as randomized through 7 days after started on designated respiratory therapy. All-cause mortality was monitorted during the entire initial hospitalization, an average of 4 months.
Description: All participants in the study were inpatients and received 24 hour care. Routine assessments such as head ultrasounds and xrays were reviewed by the research team for adverse events.
Arm/Group | Nasal High-frequency Jet Ventilation (nHFJV) | Nasal Intermittent Positive Pressure Ventilation (NIPPV)
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal High-frequency Jet Ventilation (nHFJV) (N=2) | Nasal Intermittent Positive Pressure Ventilation (NIPPV) (N=2)
Intraventricular Hemorrhage (IVH) (Nervous system disorders) | 1 (1) | 2 (2) — Very preterm infants are at high risk for developing IVH and routine head ultrasounds are done at 7-10 days. All infants were diagnosed with a grade 4 IVH but were not related to the study.
Spontaneous Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early due to concerns related to the spontaneous intestinal perforation and abdominal distension that is inherent with all forms of nasal respiratory support. There is not enough data to run statistical analysis on and there is no way to make any meaningful conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03558737/Prot_SAP_000.pdf